CLINICAL TRIAL: NCT03521908
Title: Risk of Major Bleeding Associated With Apixaban Verses Warfarin in the Treatment of Venous Thromboembolism in US Clinical Practice
Brief Title: A Study to Compare the Risk of a Major Bleeding in Participants Who Received Blood Thinning Medications Following a Blood Clot
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-523
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Venous Thromboembolism (VTE)
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants treated with apixaban
- Participants treated with warfarin

SUMMARY:
A study to compare the risk of a major bleeding in participants who received 2 different blood thinning medications following a blood clot

ELIGIBILITY:
Inclusion Criteria:

* An acute-care inpatient encounter with a principal or secondarydiagnosis of VTE, or an ambulatory-care encounter with any diagnosis of VTE
* An outpatient pharmacy claim for apixaban or warfarin during the 30-day period following the index encounter
* Continuous and comprehensive medical/drug coverage for ≥6 months preceding the index encounter

Exclusion Criteria:

* Evidence of a trial fibrillation/flutter or chemotherapy/radiation therapy for malignancy (other than non-melanoma skin cancer) during 6-month period preceding first receipt of index therapy
* Evidence of VTE(VTE event)during 6-month period preceding index encounter
* Evidence of malignancy (other than non-melanoma skin cancer) during 90-day period preceding first receipt of index therapy

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise all persons aged ≥18 years who received outpatient treatment with apixaban or warfarin within 30 days following their first observed encounter for VTE, and who met all other qualifying criteria.
Sampling Method: Probability Sample
Enrollment: 35756 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
Incidence of major bleeding in participants treated with apixaban | 2 years
Incidence of major bleeding in participants treated with warfarin | 2 years

SECONDARY OUTCOMES:
Incidence of clinically relevant non-major bleeding event in participants treated with apixaban | 2 years
Incidence of clinically relevant non-major bleeding event in participants treated with warfarin | 2 years
Incidence of recurrent VTE in participants treated with apixaban | 2 years
Incidence of recurrent VTE in participants treated with warfarin | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Princeton, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm